CLINICAL TRIAL: NCT04723875
Title: Postoperative Adjuvant Chemotherapy in Early-stage Cervical Cancer That Not Meet Criteria of Adjuvant Therapeutic According to NCCN Guideline: A Prospective Multicenter Randomized Controlled Clinical Trial
Brief Title: Postoperative Adjuvant Chemotherapy in Early-stage Cervical Cancer That Not Meet Criteria of Adjuvant Therapeutic According to NCCN Guideline
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Hunan Cancer Hospital (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Obstetrics and Gynecology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-S113
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Docetaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant chemotherapy group (Experimental): Participant will receive 3 cycles of adjuvant chemotherapy if having any of the following factors；participant will receive 6 cycles of adjuvant chemotherapy if having ≥2 of the following factors.
  Risk factors: (1) Deep cervical invasion（≥ 2/3）；（2）Differentiation grade 2-3；（3）Lymphatic vascular space infiltration；（4）Adenocarcinoma or adenosquamous carcinoma；（5）Tumor size ≥ 2cm
  Interventions: Drug: Paclitaxel or docetaxel + Cisplatin or carboplatin
- Control group (No Intervention): The participants receive no intervention.

INTERVENTIONS:
Drug: Paclitaxel or docetaxel + Cisplatin or carboplatin — Paclitaxel 135-175mg/m2 over 3 hours or docetaxel 70-75 mg/m2， 30min ＋ Cisplatin 75-80mg/m2 or carboplatin AUC = 5, repeat per 21 days.
  Arms: Adjuvant chemotherapy group

SUMMARY:
This is a prospective, phase 3 randomized controlled clinical trial. Cervical cancer patients who undergo radical surgery but do not meet criteria of adjuvant therapy according to NCCN guideline are enrolled to receive adjuvant chemotherapy. The primary endpoint was disease-free survival (DFS) rate at 3 year. The secondary endpoints were 5-year DFS, overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 2018 FIGO staged IB1, IB2, IIA1 cervical cancer.
2. The initial treatment was radical hysterectomy + pelvic lymphadenectomy by laparotomy or laparoscopy with cervical cancer foci sealed before dissection of the vagina and without uterine manipulator.
3. Postoperative pathological diagnosis was cervical squamous cell carcinoma, cervical adenosquamous cell carcinoma or cervical adenocarcinoma.
4. Assessment of risk factors not meeting Sedlis criteria （NCCN guideline），but having one of following factors ：（1）Deep stromal infiltration（≥2/3 layer）；（2）histopathological differentiation grade G2 ~ G3；（3）Lymph-vascular space invasion ；（4）Adenocarcinoma or adenosquamous cell carcinoma；（5）Tumor size ≥2cm.
5. Age：18-70 years old.
6. WBC≥3.5*10^9/L, NEU≥1.5*10^9/L, Platelet≥80×10^9 /L; AST and ALT ≤1.5 times normal upper limit; Total bilirubin ≤1.5 times the upper limit of normal value; serum creatinine and blood urea nitrogen ≤the upper limit of normal value.
7. Eastern Cooperative Oncology Group score 0-1.
8. Well-compliance and willing to keep in touch.
9. Willing to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. Postoperative pathology has high-risk factors（lymph node metastasis, parametrial infiltration or positive surgical margin）or meets Sedlis criteria.
2. Participate in other clinical trials at the same time.
3. Comorbidity including but not limited to: heart diseases (grade III-IV cardiac insufficiency (NYHA standard); central nervous system diseases or nonfunctional behavior; hematological system diseases; liver or kidney malformation or history of surgery.
4. Persons without disposing capacity.
5. Drug and/or alcohol abuse.
6. Unable or unwilling to sign informed consents.
7. Not eligible for the study judged by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 year
  DFS is defined as the time interval between the date of random assignment and the date of the first documented evidence of relapse at any site or death related to cancer (including toxicity), whichever occurred first.

SECONDARY OUTCOMES:
Overall survival （OS） | 3 year
  OS is defined as the time from the date of randomization until death of any cause.
5-year DFS/OS | 5 years
  DFS is defined as the time interval between the date of random assignment and the date of the first documented evidence of relapse at any site or death related to cancer (including toxicity), whichever occurred first. OS is defined as the time from the date of randomization until death of any cause.
Incidence of Toxicity | 2 years
  The toxicity induced by chemotherapy during observation time will be estimated on the basis of the National Cancer Institute Common Toxicity Criteria Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, M.D., PhD, Study Chair — Tongji Hospital
Locations (3):
- China (3):
  - Tongji Hospital, Wuhan, Hubei
  - Qilu Hospital, Shandong University, 107 West Wenhua Road, Ji'nan, Shandong
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang